CLINICAL TRIAL: NCT00332267
Title: Cerebral Blood Flow and Metabolism During Hypoxia and Endotoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); H:S, Denmark (Unknown); The Danish National Research Foundation, Denmark (Unknown)
Responsible Party: Kirsten Moller, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KM-HYP/ETX
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Hypoxia; Endotoxemia; Healthy
Keywords: Sepsis; Hypoxia; Altitude Sickness; Endotoxin; Cytokines; Cerebral blood flow; Cerebral metabolism; Reactive oxygen species
MeSH Terms: conditions — Hypoxia; Endotoxemia; Sepsis; Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endotoxin infusion, Normobaric hypoxia

SUMMARY:
The objective of the present protocol is to study whether a low level of oxygen in the blood will affect the immune response to as well as cerebral blood flow and metabolism during an infection and, conversely, whether the acute systemic and cerebral physiologic response to hypoxia is modified by an ongoing inflammatory response.

DETAILED DESCRIPTION:
The combination of acute infection and a low level of oxygen in the blood is a common phenomenon. Thus, acute hypoxia may complicate severe infections including severe sepsis. Conversely, healthy persons who ascend to moderately high altitudes, which will be associated with a lowering of the inspired oxygen level, may sustain an infection. Even so, it is unknown whether hypoxia modifies the systemic inflammatory response, or, conversely, whether the reaction to hypoxia is influenced by the presence of systemic inflammation. The present protocol aims to measure global cerebral blood flow, metabolism and net flux as well as the systemic response in healthy volunteers who are subjected to either normobaric hypoxia alone (N=12), low-dose IV endotoxin infusion alone (N=12), or a combination of endotoxin infusion and normobaric hypoxia (N=12).

ELIGIBILITY:
Inclusion Criteria:

* Healthy nonsmoking male
* Age 18-45 yrs

Exclusion Criteria:

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow | 0, 9 hours
Cerebral oxygen metabolism | 0, 9 hours
Plasma cytokine content | 0, 4, 19, 12 hours
Lake Louise Score | 0, 4, 9, 12 hours
ESQ-C | 0, 4, 9, 12 hours
Endotoxemia Score | 0, 4, 9, 12 hours

SECONDARY OUTCOMES:
Cerebral net flux | 0, 9 hours
Mean arterial pressure | Hourly, 0 through 12 hours
Heart rate | Hourly, 0 through 12 hours
Oxygen saturation | Hourly, 0 through 12 hours
Body temperature | Hourly, 0 through 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Taudorf, MD, Principal Investigator — Rigshospitalet, Denmark; Kirsten Moller, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center of Inflammation and Metabolism, Rigshospitalet, Copenhagen, Denmark